CLINICAL TRIAL: NCT02715297
Title: Adjuvant Stereotactic Fractionated Radiotherapy to the Resection Cavity in Recurrent Glioblastoma
Acronym: GlioCave/NOA17
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: Helmholtz Zentrum München (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RadOnc MRI TUM - 1
Record Dates: First submitted 2016-02-29; First posted 2016-03-22 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Glioblastoma
Keywords: glioblastoma; GBM; radiotherapy; Re-irradiation; progression
MeSH Terms: conditions — Glioblastoma; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: SRT to the resection cavity (Experimental): Postoperative stereotactic fractionated radiotherapy (SRT) to the resection cavity to a Total Dose of 46 Gy, 2 Gy single dose, or 36 Gy in 3 Gy single dose 5 fractions/week, depending on the volume and location of the treatment region.
  Interventions: Radiation: SRT to the resection cavity
- Arm B: Observation (No Intervention): Observation without adjuvant radiotherapy.

INTERVENTIONS:
Radiation: SRT to the resection cavity — 46 Gy total dose will be delivered in 2 Gy per fraction, or 36 Gy delivered in 3 Gy per fraction, 5 fractions within 1 week. Doses will have to cover 95% of the PTV with the prescribed dose. The clinical target volume (CTV) will be defined as the resection cavity of the recurrent glioblastoma plus a margin of 5mm. A CTV to PTV margin of 1 to 3mm will be added according to technique used for immobilisation.
  Arms: Arm A: SRT to the resection cavity

SUMMARY:
This multi-center randomized controlled phase II trial will investigate the impact of stereotactic fractionated radiotherapy to the resection cavity of complete resected recurrent glioblastoma on progression free survival. As secondary endpoints, overall survival, safety and toxicity as well as early response criteria on MRI, quality of life and neurocognitive function will be assessed. Chemotherapy will not be part of the protocol, however, additional treatment will be possible upon investigators best choice.

DETAILED DESCRIPTION:
The treatment of recurrent glioblastoma is, beside of its abundance in clinical practice, still under discussion. Patients presenting with recurrent disease are therefore treated within individual concepts, largely based on small prospective trials, retrospective evaluations or case reports. Therefore, the treatment ranges from best supportive care over primary systemic treatments towards local therapies such as radiotherapy or surgical resection. Even if there might be a large selection bias, local therapies with or without concomitant or adjuvant chemotherapy seem to promise the largest prognostic benefit. Whether the combination of surgical resection and adjuvant radiotherapy improves survival, as it does within the primary situation, is unknown.

The result of surgical resection might have an impact as well. Several case reports, retrospective evaluations and prospective studies have also included patients with remaining gross tumor after maximum save resection. In these trials, radiotherapy was associated with improvements in progression free as well as overall survival. Therefore, the influence of neuroimaging on prognosis is currently evaluated within the GLIA-A trial. Furthermore, stereotactic radiotherapy with or without an experimental systemic therapy is currently investigated within another multicenter randomized trial (NOA-12).

Whether patients might benefit from a postoperative radiotherapy of the resection cavity after complete extirpation of all macroscopic tumor is key question of this protocol.

To answer this question, the considered standard of care after complete resection, namely observation with or without adjuvant systemic therapy, will be compared to a postoperative normofractionated stereotactic radiotherapy towards the resection cavity within an open label, randomized trial. The prescribed total dose will be 46 Gy in 2 Gy fractions of 36 Gy in 3 Gy fractions depending on the treatment volume.

Concerning safety, side effects will be monitored prospectively. Safety parameters will be compared between both arms of the study. Furthermore, measures for quality of life, neurocognitive function as well as neuroimaging features will be evaluated prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Unifocal, supratentorial recurrent glioblastoma
* Prior course of standard treatment
* Complete resection of all contrast enhancing areas
* age ≥ 18 years of age
* Karnofsky Performance Score 60% or higher
* For women with childbearing potential, (and men) adequate contraception.
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* Multifocal glioblastoma of gliomatosis cerebri
* Time interval of less than 6 months after primary radiotherapy
* Previous re-irradiation or prior radiosurgery of prior treatment with interstitial radioactive seeds
* refusal of the patients to take part in the study
* Patients who have not yet recovered from acute toxicities of prior therapies
* Known carcinoma < 5 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy
* Pregnant or lactating women
* Participation in another clinical study or observation period of competing trials, respectively.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2016-02; Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) at 12 months | 1 year
  PFS will be defined according to the MacDonald and RANO-Criteria; Complete remission: Remission of all contrast-enhanced lesions on CT or MRI without worsening of neurologic status
  Partial remission: at least 50% remission of the contrast-enhancing lesions on CT or MRI without increase in steroid medication and without worsening of the neurologic status
  Stable disease: Remission of the solid tumor/contrast-enhancing lesion on CT or MRI of less than 50% or progression of the solid tumor/contrast-enhancing lesion on CT or MRI of less than 25%, without increase in steroid medication of worsening of the neurologic status
  Progression: Increase in solid tumor/contrast-enhancing lesion of 25% or more or development of a new lesion

SECONDARY OUTCOMES:
Overall survival | 1 year
  Patients will be followed up until death or for at least 1 year. Living patients will be censored according to the date of their last visit.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 1 year
  Safety and tolerability will be assessed by quality and quantity according to the International Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 for toxicity and adverse event reporting. Safety and toxicity of the study treatment will be evaluated by clinical neurological examination as well as neuro-imaging studies (MRI or CT).
Quality of Life questionnaire | 1 year
  The EORTC QLQ-C30 version 3.0 questionnaire will be used to monitor for Quality of Life continuously throughout the treatment course as well as during follow up.
Neurocognitive function | 1 year
  Neurocognitive function will be assessed at randomisation, at 6 months and at 12 months after randomization. A battery containing of 3 tests will be used. For assessment of learning, early and intermediate recall, the German version of the California Verbal Learning Test (CVLT) as well as the Regensburger Wortflüssigkeits-Test (RWT) will be used. Cognitive flexibility, speed as well as attention will be tested by the Trail-Making-Test. The tests at 6 and at 12 months will be compared to the result of the baseline measure as well as to each other.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie E. Combs, Prof. Dr., Principal Investigator — Klinik für RadioOnkologie und Strahlentherapie
Locations (1):
- Dept. Radiation Oncology, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Straube C, Scherb H, Gempt J, Kirschke J, Zimmer C, Schmidt-Graf F, Meyer B, Combs SE. Adjuvant stereotactic fractionated radiotherapy to the resection cavity in recurrent glioblastoma - the GlioCave study (NOA 17 - ARO 2016/3 - DKTK ROG trial). BMC Cancer. 2018 Jan 3;18(1):15. doi: 10.1186/s12885-017-3928-7. PMID 29298660